CLINICAL TRIAL: NCT06773624
Title: Evaluation of 68Ga-DOTATOC PET/CT-enterography for the Detection of the Primary Lesion in Neuroendocrine Tumors of the Small Bowel
Brief Title: Use of 68Ga-DOTATOC PET/CT-enterography for Detection of the Primary Lesion in Neuroendocrine Tumors of the Small Bowel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 1441
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Small Bowel Neoplasia; Neuroendocrine (NE) Tumors
MeSH Terms: conditions — Neoplasms | interventions — Ga(III)-DOTATOC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET/CT-enterography with 68Ga-DOTATOC (Other): Patients underwent to PET/CT-enterography with 68Ga-DOTATOC
  Interventions: Other: PET/CT-enterography with 68Ga-DOTATOC

INTERVENTIONS:
Other: PET/CT-enterography with 68Ga-DOTATOC — Patients underwent to PET/CT-enterography with 68Ga-DOTATOC

SUMMARY:
The neuroendocrine neoplasms of the small intestine (Si-NENs) is a relatively rare malignancy. Surgical resection is the only curative treatment for the early-stage. It remains controversial its application for advanced metastatic gastroenteropancreatic neuroendocrine tumours (GEP-NETs).

The identification of metastatic disease and tumor grade are the most important prognostic factors in advanced GEPNETs. Therefore, precise staging and evaluation of disease burden with a reliable imaging method is crucial for determining the correct stage of the disease and consequently the correct treatment.

A unique feature of NeuroEndocrinal Tumors (NETs) is the expression of somatostatin receptors (SSTR) which can be targeted with radiolabeled peptides for imaging.

The Positron Emission Tomography-Computed Tomography (PET/CT) technique using somatostatin analogs labeled with the positron emitting isotope, 68Ga (68Ga-DOTA peptides), has been shown to offer advantages over conventional imaging modalities as well as additional important quantitative and qualitative diagnostic information.

The aim of this study is to calculate the sensitivity (SE), the specificity (SP), the positive and negative predictive values (PPV and NPV) and the overall accuracy of 68Ga-DOTATOC PET/CT-enterography in detecting in primary lesion and multifocality of siNETs.

ELIGIBILITY:
Inclusion Criteria:

* patients with small bowel neuroendocrine tumours
* tumors with any grade (from 1 to 3) and any Ki 67 percentage
* patients eligible for surgical resection

Exclusion Criteria:

* patients with synchronous other oncological disease
* patients with Inflammatory bowel disease
* patients Not eligible for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of predictive role of CT-Enterography and 68Ga-DOTATOC PET/CT in detecting siNETs | 3 months
  Proportion of the true positive patients at diagnostic procedure considering the pathology results as the gold standard.

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No